CLINICAL TRIAL: NCT00287235
Title: A Prospective, Controlled Study Of The Clinical Efficacy Of Albumin Dialysis Using The Molecular Adsorbent Recirculating System (MARS®) For The Treatment Of Patients With Hepatic Encephalopathy
Brief Title: Efficacy of Albumin Dialysis to Treat Patients With Hepatic Encephalopathy Using The Molecular Adsorbent Recirculating System (MARS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Gambro Renal Products, Inc. (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MARS HE Study
Record Dates: First submitted 2006-02-02; First posted 2006-02-06 (Estimated); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Hepatic Encephalopathy; Liver Failure; Hepatitis, Chronic; Liver Cirrhosis
Keywords: Hepatic Encephalopathy; End Stage Liver Disease; Cirrhosis; MARS; Albumin Dialysis
MeSH Terms: conditions — Hepatic Encephalopathy; Liver Failure; Hepatitis, Chronic; Liver Cirrhosis; End Stage Liver Disease; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Standard Medical Therapy + MARS (Experimental): Patients who were randomized to Group 1 received daily MARS treatments in addition to Standard Medical Therapy for 5 consecutive days.
  Interventions: Device: MARS; Drug: Standard Medical Therapy
- Group 2: Standard Medical Therapy Only (Active Comparator): Patients who were randomized to Group 2 received standard medical treatment only.
  Interventions: Drug: Standard Medical Therapy

INTERVENTIONS:
Device: MARS
  Other Names: ECAD; Extracorporeal Albumin Dialysis
  Arms: Group 1: Standard Medical Therapy + MARS
Drug: Standard Medical Therapy
  Other Names: SMT

SUMMARY:
The primary objective of the study was to compare the efficacy, safety and tolerability of Extracorporeal Albumin Dialysis (ECAD) using the Molecular Adsorbent Recirculating System (MARS®) device in improving severe HE by 2 grades compared to Standard Medical Therapy (SMT) in patients with chronic End Stage Liver Disease (ESLD) during a 5 day study period.

DETAILED DESCRIPTION:
The trial was a two-group unblinded multicenter clinical trial. Patients were randomized to receive either SMT or SMT plus five days MARS® treatment. The trial design called for patients to receive a baseline hepatic encephalopathy (HE) assessment on admission, and at 12-hour intervals, giving 10 HE measurements during treatment using a refinement / adaptation of the Conn West Haven HE Criteria HE scoring system

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent by patient or patient's legally appointed representative
2. Be at least 18 years of age; male or female
3. Have chronic end stage liver disease with worsening Hepatic Encephalopathy (Grades 3,4).

Exclusion Criteria:

1. Clinically significant bleeding from gastrointestinal or other site within the last 24 hours and requires 2 or more units of blood to maintain a stable hemoglobin level
2. Hemodynamically unstable or on vasopressor agents for blood pressure support (except for renal-dosed dopamine)
3. On acute or chronic hemodialysis or continuous renal replacement therapy (CRRT)
4. Pregnancy
5. Inability to obtain informed consent
6. Uncontrolled sepsis as defined by hemodynamic instability
7. Post-liver transplant
8. Fulminant hepatic failure
9. Irreversible brain damage as indicated by the neurologic examination and CT imaging
10. Endocarditis
11. Pulmonary edema
12. Massive aspiration pneumonia secondary to Hepatic Encephalopathy
13. Active alcohol consumption as determined by a positive blood ethanol level on enrollment/admission
14. Acute main portal vein thrombosis in patients with Hepatocellular Carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2000-09; Primary Completion 2003-11 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Two-point reduction in HE score from the randomization grade | Within the five-day treatment period
  The primary outcome measure was a two-point reduction in HE score from the the randomization grade (i.e. Grade 4 improved to at least Grade 2 and Grade 3 improved to at least Grade 1). Two summary statistics were used in the analysis: 1) The proportion of HE readings within the five-day treatment period showing an improvement of at least two points over baseline 2) The time from admission to the first two-point improvement in HE score.

SECONDARY OUTCOMES:
Magnitude, duration and time of improvement in Hepatic Encephalopathy | Within the five-day treatment period
Cognitive function and functional status of patients | Within the five-day treatment period
Renal function, serum bilirubin, bile acids, prothrombin activity and the hemodynamics of patients with Hepatic Encephalopathy | Within the five-day treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Hassanein, MD, Principal Investigator — University of California San Diego Medical Center (UCSD)
Locations (8):
- United States (6):
  - University of Alabama, Birmingham, Alabama
  - University of California, San Diego, San Diego, California
  - Northwestern University, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Columbia-Presbyterian Medical Center, New York, New York
  - University of Virginia, Charlottesville, Virginia
- UZ Gasthuisberg, Leuven, Belgium
- University Hospital of Copenhagen, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Result] Hassanein TI, Tofteng F, Brown RS Jr, McGuire B, Lynch P, Mehta R, Larsen FS, Gornbein J, Stange J, Blei AT. Randomized controlled study of extracorporeal albumin dialysis for hepatic encephalopathy in advanced cirrhosis. Hepatology. 2007 Dec;46(6):1853-62. doi: 10.1002/hep.21930. PMID 17975845